CLINICAL TRIAL: NCT04218461
Title: Evaluation of the Usability of the Delirium Prediction Model of PRE-DELIRIC (PREdiction of DELIRium) in Medical ICU Patients
Brief Title: PREdiction of DELIRium in Medical ICU Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Assistant Professor, Istanbul Demiroglu Bilim University
Other Study IDs: 2019-08
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Delirium; Intensive Care Unit Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PRE-DELIRIC model — To predict delirium according to risk factors in the PRE-DELIRIC model

SUMMARY:
In intensive care unit (ICU) patients, the ability to predict delirium may help reduce its incidence, duration, and severity. The PREdiction of DELIRium in ICU (PRE-DELIRIC) model was recently developed for this purpose. Our aim was to test the PRE-DELIRIC model in the medical ICU.

DETAILED DESCRIPTION:
Delirium, a disturbance of consciousness with an acute onset and a variable course of impaired cognitive functioning, is common in patients admitted to the ICU. Several tools are available for assessing delirium in ICU patients, of which the confusion assessment method-intensive care unit (CAM-ICU) has the highest sensitivity and specificity.

Although several predictive models for non-intensive care patients exist, as well as one for older medical intensive care patients, no evidence based prediction model for general intensive care patients is available. Also the tools are not involved the metabolic parameters which cause delirium. Because of that the tool need to have biochemical parameters.

In the light of these information our aim is to validate the PRE-DELIRIC model in medical ICU in Turkish people.

ELIGIBILITY:
Inclusion Criteria:

* be at the medical ICU
* 18 and older years of age
* predict to stay in the ICU over 24 hours
* not to be pregnant
* not to be breastfeeding
* not to have dementia, alcoholism
* have not previously received a diagnosis of delirium
* have not communication problem
* agree to participate to the study by patient's relatives

Exclusion Criteria:

* younger than 18 years old
* stay in the ICU less than 24 hours
* be pregnant
* breastfeeding
* have dementia, alcoholism
* previously received a diagnosis of delirium
* have communication problem
* not agree to participate to the study by patient's relatives

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stay in the medical ICU
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Predict of delirium risk with questionnare | up to 20 weeks
  CAM-ICU will be used for defining the delirium risk. We define delirium as a minimum of one positive CAM-ICU screening during each patient's intensive care stay developed and validated for ICU patients, assesses 10 risk factors for delirium that are readily observable within the first 24 hours following ICU admission. CAM-ICU scale includes of four items. The items are about level of consciousness, assessment of attention, state of thought organization and following a simple command. In order to be diagnosed with delirium, the first two items and one of the third or fourth item must be in favor of delirium.
Predict of delirium risk with questionnare 2 | up to 20 weeks
  The PRE-DELIRIC model will be used for defining the delirium risk. The PRE-DELIRIC model developed and validated for ICU patients, assesses 10 risk factors for delirium that are readily observable within the first 24 hours following ICU admission. The model consists of biochemical parameters, used drugs, infection status.
Comparison of delirium risk with two questionnares | up to 20 weeks
  The investigator will assess the CAM-ICU and PRE-DELIRIC in the first 24 hours after the patient comes to the ICU. The PRE-DELIRIC model and CAM-ICU will use for defining the deliirum risk. The investigators will do validity and reliability of PRE-DELIRIC model in medical ICU patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten OZEN, Principal Investigator — Istanbul Demiroglu Bilim University
Locations (1):
- Demiroglu Bİlim University, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Boogaard M, Pickkers P, Slooter AJ, Kuiper MA, Spronk PE, van der Voort PH, van der Hoeven JG, Donders R, van Achterberg T, Schoonhoven L. Development and validation of PRE-DELIRIC (PREdiction of DELIRium in ICu patients) delirium prediction model for intensive care patients: observational multicentre study. BMJ. 2012 Feb 9;344:e420. doi: 10.1136/bmj.e420. PMID 22323509
- [Background] Sosa FA, Roberti J, Franco MT, Kleinert MM, Patron AR, Osatnik J. Assessment of delirium using the PRE-DELIRIC model in an intensive care unit in Argentina. Rev Bras Ter Intensiva. 2018 Mar;30(1):50-56. doi: 10.5935/0103-507x.20180010. PMID 29742219
- [Background] Green C, Bonavia W, Toh C, Tiruvoipati R. Prediction of ICU Delirium: Validation of Current Delirium Predictive Models in Routine Clinical Practice. Crit Care Med. 2019 Mar;47(3):428-435. doi: 10.1097/CCM.0000000000003577. PMID 30507844